CLINICAL TRIAL: NCT03823222
Title: Proteins From Duckweed Trial
Acronym: ProDuckT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Diederik Esser, project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL66859.081.18
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Degree of Digestilbility
Keywords: Duckweed protein; protein; degree of digestibility; whey protein
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duckweed protein (Experimental): 20 gram of isolated protein
  Interventions: Dietary Supplement: Duckweed protein
- Whey protein (Experimental): 20 gram of isolated protein
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Duckweed protein — 20 grams isolated protein
  Arms: Duckweed protein
Dietary Supplement: Whey protein — 20 grams isolated protein
  Arms: Whey protein

SUMMARY:
This study aims to study the digestibility of isolated duckweed protein. The digestibility of the isolated duckweed protein will be compared to an isolated benchmark protein whey.

Objective: The primary objective is to investigate the digestibility of isolated duckweed protein and the isolated benchmark protein whey.

Study design: The study is a cross-over, double blind, controlled trial in which study participants will visit the research facility on two occasions under fasting conditions. Subjects will receive two protein sources in randomized order with a washout period of one week. Blood will be collected via a catheter before and up-to 3 hours after protein consumption.

Study population: We aim to include 12 healthy volunteers aged 18-50 years. Intervention: Study participants will receive 20 grams of isolated duckweed protein and the isolated benchmark protein whey.

Main study parameters/endpoints: The main study parameter is blood amino acids measured before and after consumption of 20 g protein.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 25 kg/m2
* Having veins suitable for blood sampling via a catheter (judged by study nurse/ medical doctor)

Exclusion Criteria:

* Any metabolic, gastrointestinal, inflammatory or chronic disease (such as diabetes, anaemia, hepatitis, cardiovascular disease)
* History of gastro-intestinal surgery or having (serious) gastro-intestinal complaints
* History of liver dysfunction (cirrhosis, hepatitis) or liver surgery
* Kidney dysfunction (self-reported)
* Use of medication that may influence the study results, such as gastric acid inhibitors, laxatives, stomach protectors and drugs that can affect intestinal motility
* Anaemia (Hb values <7.5 for women and <8.5 for men)
* Reported slimming, medically prescribed, vegan/vegetarian or other extreme diets or the use of protein supplements
* Not willing to give up blood donation during the study
* Current smokers
* Alcohol intake ≥4 glasses of alcoholic beverages per day
* Pregnant, lactating or wishing to become pregnant in the period of the study (self-reported)
* Abuse of illicit drugs
* Food allergies for products that we use in the study
* Participation in another clinical trial at the same time
* Being an employee of the department Consumer Science & Health group of Wageningen Food & Biobased Research

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Change in blood free amino acids (e.g. Degree of digestibility) | 20 gram protein will be consumed and blood samples will be taken before and up to 3 hours after protein consumption
  postprandial test, determine free amino acids in blood samples collected before and after a postprandial challenge test

SECONDARY OUTCOMES:
change in plasma insulin | 20 gram protein will be consumed and blood samples will be taken before and up to 3 hours after protein consumption
  before and after a postprandial challenge test
change in plasma glucose | 20 gram protein will be consumed and blood samples will be taken before and up to 3 hours after protein consumption
  before and after a postprandial challenge test

OTHER OUTCOMES:
change in visual analogue scale (VAS) scores on intestinal complains | daily from day1 until day3 after the intervention
  On a scale ranging from worst-best outcome (higher scores are better)

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Esser, PhD, Principal Investigator — Wageningen Research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
will not be shared